CLINICAL TRIAL: NCT07319832
Title: A Multicenter, Retrospective and Prospective, Observational Study to Evaluate the Efficacy and Safety of Subcutaneous Teduglutide in the Treatment of Short Bowel Syndrome (SBS) in Parenteral Nutrition (PN) Dependent Chinese Pediatric Subjects (≥1 Through 17 Years Old)
Brief Title: A Study of Teduglutide in Chinese Children and Teenagers With Short Bowel Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-633-5002
Record Dates: First submitted 2025-12-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Short Bowel Syndrome (SBS)
Keywords: Drug Therapy
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Retrospective Group: Participants who completed the 24-week teduglutide treatment period before enrollment will have their clinical data collected retrospectively from their medical records.
  Interventions: Other: No Intervention
- Mixed Group: Participants who initiated treatment before the study start date but have not completed the 24-week teduglutide treatment period at the time of enrollment will have their clinical data collected retrospectively before enrollment and prospectively after enrollment.
  Interventions: Other: No Intervention
- Prospective Group: Participants who will initiate the teduglutide treatment period after enrollment will have their clinical data collected prospectively for 48 weeks.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
Short Bowel Syndrome (SBS) is a rare condition that happens when a large part of the bowel (also called intestine) is missing or has been removed because of illness or surgery. In children, SBS means that the intestine cannot absorb enough food, water and important part of food the body needs (called nutrients) because a big part of it has been removed, bypassed or did not develop normally at birth and the children need support through a vein (parenteral support or PS) for more than 42 days to stay healthy and keep their energy. SBS in children is defined mainly by how well the intestine works and how long the children need this support, not just by how long the intestine is.

The main aim of the study is to learn how well the teduglutide works in children and teenagers with SBS and who need PS. Another aim is to find out how well teduglutide works for participants to lower the amount of PS needed. Also, the study wants to learn more about how safe teduglutide is in children and teenagers with SBS who need PS.

The study will review data already existing in the medical records of participants as well as collect new data during the study.

ELIGIBILITY:
Inclusion criteria

* Children and adolescents greater than or equal to (>=)1 through 17 years of age at Day 1 (D1).
* Documented diagnosis of SBS.
* Received or plan to receive Teduglutide treatment for a minimum of 24 weeks.
* Stable PN/IV support, defined as inability to significantly reduce PN/IV support, usually associated with minimal or no advance in enteral feeds (i.e., 10% or less change in PN or advance in feeds) for at least 3 months prior to D1, as assessed by the investigator. Transient instability for events such as interruption of central access or treatment for sepsis is allowed if the PN/IV support returns to within 10% of baseline prior to the event.
* Informed consent obtained from the patient aged 8 to 17 years and their guardians, while informed consent from the guardians for participants under 8 years old, unless waived by the Institution's Ethics Committee.

Exclusion criteria

* Participants who are not expected to be able to advance oral or tube feeding regimens.
* Serial Transverse Enteroplasty (STEP) or any other bowel lengthening procedure performed within 3 months prior to baseline.
* Known clinically significant untreated intestinal obstruction contributing to feeding intolerance and inability to reduce PS.
* Evidence of clinically significant obstruction on upper GI series done within 6 months prior to baseline.
* Previous use of octreotide or Dipeptidyl peptidase-4 (DPP-4) inhibitors within 3 months prior to baseline.
* Signs of active, severe, or unstable clinically significant hepatic impairment during the screening or baseline period, indicative by any of the following laboratory test results:

  1. Total Bilirubin Level (TBL) >= 2 × upper limit of normal (ULN)
  2. Aspartate Aminotransferase (AST) >=7 × ULN
  3. Alanine Aminotransferase (ALT) >=7 × ULN

     For Participants with Gilbert's disease:
  4. Indirect (unconjugated) bilirubin >=2 × ULN
* Signs of known continuous active or unstable, clinically significant renal dysfunction shown by results of an estimated glomerular filtration rate (eGFR) below 50 millilitres per minutes per 1.73 meter square (mL/min/1.73 m^2).
* Known hypersensitivity of the active substance or excipient of teduglutide.
* Body weight less than (<) 10 kg at baseline.
* Previous use of teduglutide or native/synthetic Glucagon-like Peptide-2 (GLP-2).
* Previous use of GLP-1 analog or human growth hormone within 3 months prior to baseline.
* Any condition, disease, illness, or circumstance that in the investigator's opinion puts the patient at any undue risk, prevents completion of the study, or interferes with analysis of the study results.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consists of Chinese pediatric participants with SBS who are dependent on PS.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Who Achieve at Least a 20% Reduction from Baseline in Weekly Parenteral Support (PS) Volume at Week 24 | At Week 24
  Percentage of participants who achieve at least a 20 percent (%) reduction from baseline in weekly PS volume at Week 24 will be reported.

SECONDARY OUTCOMES:
Number of Participants Able to Completely Wean off PS Support at Week 24 | At Week 24
  Number of participants who are able to completely wean off PS support at Week 24 will be reported.
Absolute Change from Baseline in PN/Intravenous (IV) Support Volume | Baseline up to Week 24
  Absolute change from baseline in PN/IV support volume will be reported.
Percent Change From Baseline in PN/IV Support Volume | Baseline up to Week 24
  Percent change from baseline in PN/IV support volume will be reported.
Absolute Change From Baseline in PN/IV Support Calories | Baseline up to Week 24
  Absolute change from baseline in PN/IV support calories will be reported.
Percent Change From Baseline in PN/IV Support Calories | Baseline up to Week 24
  Percent change from baseline in PN/IV support calories will be reported.
Absolute Change From Baseline in Plasma Citrulline | Baseline, Week 24
  Absolute change from baseline in plasma citrulline will be reported.
Percent Change From Baseline in Plasma Citrulline | Baseline, Week 24
  Percent change from baseline in plasma citrulline will be reported.
Absolute Change From Baseline in Enteral Nutrition (EN) Support Volume | Baseline up to Week 24
  Absolute change from baseline in EN support volume will be reported.
Percent Change From Baseline in EN Support Volume | Baseline up to Week 24
  Percent change from baseline in EN support volume will be reported.
Absolute Change From Baseline in EN Support Calories | Baseline up to Week 24
  Absolute change from baseline in EN support calories will be reported.
Percent Change From Baseline in EN Support Calories | Baseline up to Week 24
  Percent change from baseline in EN support calories will be reported.
Change From Baseline in Hours per day of PN/IV Support | Baseline up to Week 24
  Change from baseline in hours per day of PN/IV support will be reported.
Change From Baseline in Days per Week of PN/IV Support | Baseline up to Week 24
  Change from baseline in days per week of PN/IV support will be reported.
Percentage of Participants with at Least a 20% Reduction From Baseline in PN/IV Volume | Baseline up to Week 24
  Percentage of participants with at least a 20% reduction from baseline in PN/IV volume will be reported.
Change in Body Weight | Baseline up to Week 24
  Change in body weight will be reported.
Change in Height | Baseline up to Week 24
  Change in height will be reported.
Change in Head Circumference | Baseline up to Week 24
  Head circumference will be measured in participants 36 months of age and younger.
Change in Height Z-score | Baseline up to Week 24
  Height is measured using Z-score. Z score is calculated as ([observed value/M]^L-1)/S*L, where observed value is the child's height. The L, M, and S values vary according to the child's sex and age.
Change in Weight Z-score | Baseline up to Week 24
  Weight is measured using Z-score. Z score is calculated as ([observed value/M]^L-1)/S*L, where observed value is the child's weight. The L, M, and S values vary according to the child's sex and age.
Change in Body Mass Index (BMI) | Baseline up to Week 24
  BMI is a simple measure that uses a participant's weight and height to estimate whether they are underweight, normal weight, overweight, or obese. It is calculated as weight in kilograms (kg) divided by height in meters squared (kg/m^2). Change in BMI will be reported.
Change in BMI Z-score | Baseline up to Week 24
  BMI is measured using Z-score. Z score is calculated as ([observed value/M]^L-1)/S*L, where observed value is the child's BMI. The L, M, and S values vary according to the child's sex and age.
Number of Participants with Adverse Events (AEs). Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs) | Up to 50 weeks
  An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product. An AE does not necessarily have a causal relationship withthis treatment. An AE can therefore be any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product (investigational or marketed), whether or not considered related to treatment with the medicinal product. SAE is any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of hospitalization, results in persistent or significant disability/incapacity, results in a congenital abnormality/birth defect, or is an important medical event. An AESI is an AE (serious or nonserious) of scientific and medical concern specific to the product or program.
Number of Participants with Clinically Significant Change in Vital Sign Values | Up to 24 weeks
  Vital signs will include measurement of temperature, heart rate, blood pressure and respiratory rate. Any clinically significant change in vital signs will be determined at the investigator's discretion.
Body Weight in Participants Dependent on PS | Baseline up to Week 24
  Body weight in kg will be collected and reported.
Head Circumference in Participants Dependent on PS | Baseline up to Week 24
  Head circumference in participants 36 months of age and younger will be collected and reported.
Height in Participants Dependent on PS | Baseline up to Week 24
  Height in centimeters (cm) will be collected and reported.
Trends on Growth Chart | Baseline up to Week 24
  Trends on growth chart will be collected and reported.
Urine Output Determined up to Week 24 | Baseline up to Week 24
  Collected and calculated values of urine output will be recorded over a 48-hour period of PN/IV and EN stability before every clinic visit and within 1 week of implementing a change in the PN/IV prescription.
Fecal Output Measured by Volume | Baseline up to Week 24
  Collected and calculated values of fecal output should be recorded over a 48-hour period of PN/IV and EN stability before every clinic visit and within 1 week of implementing a change in the PN/IV prescription.
Fecal Output Measured by Number of Bowel Movements per Day | Baseline up to Week 24
  Fecal output should be recorded over a 48-hour period of PN/IV and EN stability before every clinic visit and within 1 week of implementing a change in the PN/IV prescription.
Number of Participants with Gastrointestinal-specific Testing | Baseline up to Week 24
  Gastrointestinal-specific testing will include colonoscopy or sigmoidoscopy or upper gastrointestinal (GI) endoscopy, abdominal ultrasound, fecal occult blood testing (FOBT), upper gastrointestinal series small bowel follow-through (UGI SBFT).
Number of Participants With Clinically Significant Changes in Physical Examinations | Up to 24 weeks
  Physical examination will include assessing the participants physical status. (general surface, skin, head and neck, chest [heart, lungs, breasts], abdomen [gastrointestinal, liver and gallbladder], back, urinary system, limbs, nervous system, lymph nodes, etc.). Any clinically significant change in physical examination will be determined at the investigator's discretion.
Number of Participants With Clinically Significant Changes in Laboratory Values | Up to 24 weeks
  Laboratory parameters will include hematology, chemistry and urinalysis. Any clinically significant change in laboratory values will be determined at the investigator's discretion.
Number of Participants With Clinically Significant Changes in 12-Lead Electrocardiogram (ECG) Parameters | Up to 24 weeks
  The 12-lead ECG will be evaluated. Any clinically significant change in ECG assessment will be determined at the investigator's discretion.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (4):
- China (4):
  - Guangzhou Women And Children's Medical Center, Guangzhou, Guangdong
  - Shanghai Children's Hospital, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Children's Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/